CLINICAL TRIAL: NCT06951217
Title: A Multinational, Long-Term, Safety and Tolerability, Open-Label Extension Study of Subjects Who Have Participated in Avalyn Pharma Studies of Inhaled Antifibrotic Agents (AP-LTE-008 [SAIL])
Brief Title: An Extension Study of Subjects Who Received an Avalyn Inhaled Antifibrotic Agent (SAIL)
Acronym: SAIL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Avalyn Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP-LTE-008; ACTRN12625000246482 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2025-04-08; First posted 2025-04-30 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Progressive Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Open-label AP01 treatment arm (Experimental): All trial participants will enroll from a Sponsor-led parent study of AP01 and receive open-label AP01 for continued evaluation of long-term safety and tolerability.
  Interventions: Combination Product: AP01

INTERVENTIONS:
Combination Product: AP01 — AP01 will be administered open-label via the eFlow Nebulizer System

SUMMARY:
This is an open-label extension study for participants who were previously enrolled in and completed an Avalyn Pharma Sponsored study with an inhaled antifibrotic, such as AP01. Eligible participants will have their final dose of drug at the end of study visit from the lead-in study and first AP-LTE-008 study visit on the same day.

All participants will receive 100 mg inhaled pirfenidone inhalation solution (AP01) taken twice daily using the eFlow Nebulizer System for until such a time that the drug is approved, the participant withdraws from the study, or the study is terminated.

New patients will be trained to use the nebuliser at the first treatment visit. All patients will use the eFlow nebuliser to administer AP01. Hands on training for use and cleaning of the eFlow nebuliser will be performed by site personnel with patients using the study specific instructions for use and quick reference guide provided. The first treatment for new patients will be overseen by clinic personnel.

A paper dosing diary will be used to monitor adherence along with returns of any unused investigational product.

ELIGIBILITY:
Inclusion Criteria:

* Previously participated in an Avalyn-sponsored inhaled antifibrotic clinical study for subjects with either idiopathic pulmonary fibrosis (IPF) (IPF subjects are excluded from the US and Canada) or progressive pulmonary fibrosis (PPF) and with the approval of the Study Physician.

Previous participation is defined as: Having completed the final visit of the Treatment Period on the full dose of study drug (either active or placebo).

* Male subjects and female subjects of childbearing potential (FOCBP) agree to use highly effective contraception measures from the time of first dose of study drug (for the male subject) or the signing of the informed consent form (ICF) (for the female subject), during the study, and until 90 days after the last dose of study drug. Subjects agree not to donate eggs or sperm during the same period.

Exclusion Criteria:

* Have not previously participated in an Avalyn-sponsored inhaled antifibrotic lead-in study or if the subject was permanently discontinued from the lead-in study for any reason. Subjects who discontinued study drug but continued to attend study visits are ineligible.
* Subjects who experienced an exacerbation of asthma or of chronic obstructive pulmonary disease (COPD) requiring oral or systemic corticosteroids within 3 months of Day 1 (Screening/Baseline Visit).
* Subjects who experienced an acute exacerbation of IPF (IPF subjects are excluded from the US and Canada) or of PPF within 3 months of Day 1 (Screening/Baseline Visit).
* Participation in a concurrent clinical study or in a clinical study in which any other investigational drug product aside from the Avalyn nebulized antifibrotic medication from their lead-in study was administered within the previous 30 days, or 5 half-lives of the previously administered investigational product, whichever is shorter. Subjects may be enrolled in registries.
* History of hypersensitivity and/or allergic reaction to pirfenidone or the excipients to be used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long-term safety and tolerability outcomes of subjects receiving Avalyn nebulized antifibrotic medications (AP01). | Through end of study; average of 6 years
  The incidence of adverse events will be evaluated from the time of signing of the informed consent until approximately 2 weeks after the last dose of study drug. Examples of potential adverse events include: respiratory symptoms, liver toxicity, and skin conditions. Study participants will be monitored for adverse events via the following: vital signs (blood pressure assessed using a sphygmomanometer, temperature assessed by thermometer, pulse and respiratory rate assessed by pulse oximeter), oxygen saturation, spirometry, physical exams, blood chemistry, and quality of life assessments.

SECONDARY OUTCOMES:
To evaluate the long-term effect of Avalyn nebulized antifibrotic medications on lung function the change from baseline in forced vital capacity (FVC) will be evaluated. | Through end of study; average of 6 years
  FVC will be evaluated via spirometry.
To evaluate the long-term effect of Avalyn nebulized antifibrotic medications on stabilization of disease. | Through end of study; average of 6 years
  Stabilization of disease will be based on computational analysis of quantitative high-resolution computed tomography (HRCT) to assess the extent and pattern of interstitial lung disease present on the HRCT scans (methodologies developed by Qureight).
To evaluate the long-term impact of Avalyn nebulized antifibrotic medications on subject-reported quality of life (QoL). | Through end of study; average of 6 years
  This outcome will evaluate the change from baseline in the 'Living with Pulmonary Fibrosis Symptoms and Impact Questionnaire' (L-PF) total score. The L-PF is a 23-point questionnaire with lower scores equating to 'less symptomatic' and higher scores equating to 'more symptomatic.'

CONTACTS AND LOCATIONS:
Locations (26):
- United States (9):
  - University of Colorado, Anschutz Medical Campus, Aurora, Colorado
  - Renstar Medical Research, Ocala, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Columbia University, New York, New York
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The University of Kansas Medical Center, Kansas, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
- Australia (8):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Prince Alfred Hospital, Camperdown
  - The Prince Charles Hospital (TPCH), Chermside
  - Lung & Sleep Victoria, Footscray
  - Respiratory Clinical Trials PTY Ltd, Kent Town
  - Nepean Lung & Sleep, Kingston
  - Univ of Western Australia / Institute for Respiratory Health, Nedlands
  - John Hunter Hospital, New Lambton Heights
- Canada (3):
  - Dynamic Drug Advancement, Ajax, Ontario
  - CIC Mauricie, Trois-Rivières, Quebec
  - Centre for Lung Health, Vancouver, Vancouver
- Fakultni Thomayerove nemocnice, Praha Klanovice, Czechia
- St Antonius Hospital, Nieuwegein, Netherlands
- New Zealand (2):
  - Greenlane Clinical Centre, Auckland, Auckland
  - Waikato Hospital, Hamilton
- Hospital Gregorio Marañon, Madrid, Madrid, Spain
- Leicester Biomedical Research Centre, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No